CLINICAL TRIAL: NCT04821596
Title: Study of the Mechanisms of Action of Cladribine in Multiple Sclerosis
Acronym: Clad'Action
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018/0408/HP
Record Dates: First submitted 2020-12-29; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2020-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple Sclerosis Patients (Experimental): Multiple Sclerosis Patients usually followed by Dr. Bourre as part of his consultation at the Rouen University Hospital will be offered the opportunity to participate in this study if they meet the selection criteria.
  Interventions: Other: biological collection

INTERVENTIONS:
Other: biological collection — Six 5 mL heparinized tubes, approximately 24 mL of blood will be collected as per standard practice. The 5 tubes collected from a given individual will be transported directly to the laboratory. In the laboratory, peripheral blood mononuclear cells (PBMC) will be prepared for the various analyses.
  However, in order to minimize the effect of agents other than CoA in MS patients, it is necessary that peripheral blood mononuclear cells are collected before treatment is given: for RR MS patients treated with first-line drugs (IFNβ, glatiramer acetate, teriflunomide and dimethyl fumarate, ...), RR MS patients treated with second-line drugs (natalizumab and fingolimod, ...) and RR MS patients treated with third-line drugs (alemtuzumab, ...).

SUMMARY:
The main objective of the project is therefore to study and thus better understand the immunomodulatory / anti-inflammatory effects of cladribine during multiple sclerosis.

Most current and developing therapies targeting the immune system have no effect on the progressive phase of MS, during which neurodegeneration plays a predominant role. As mentioned above, the very promising results of clinical trials with cladribine tablets for the early and progressive phase of the disease have revealed immunomodulatory properties and suggested potential neuroprotective effects.

It therefore plans to further dissect one of these two parameters by designing in vitro studies with peripheral blood mononuclear cells (PBMC) from healthy donors and MS patients.

DETAILED DESCRIPTION:
Recent clinical trials have reported a remarkable therapeutic efficacy of cladribine tablets not only in the early and recurrent phases of the disease, but also in progressive multiple sclerosis. However, its role on the immune and nervous systems has hardly been studied, although these studies suggest that CoA may exert anti-inflammatory and neuroprotective actions. Thus, the objective is to better understand/describe how cladribine acts during MS and to demonstrate whether CoA: (1) is able to effectively modulate pro-inflammatory immune processes and (2) has powerful neuroprotective properties. Ultimately, it will provide proof of concept that cladribine can be used not only in the early but also in the progressive phase of MS.

To address this hypothesis, the goal is to study the beneficial immunomodulatory/anti-inflammatory effects of cladribine on multiple sclerosis.

The main objective of this project is therefore to study and thus better understand the immunomodulatory / anti-inflammatory effects of cladribine during multiple sclerosis.

Most current and developing therapies targeting the immune system have no effect on the progressive phase of MS, during which neurodegeneration plays a predominant role. As mentioned above, the very promising results of clinical trials with cladribine tablets for the early and progressive phase of the disease have revealed immunomodulatory properties and suggested potential neuroprotective effects.

It therefore plans to further dissect one of these two parameters by designing in vitro studies with peripheral blood mononuclear cells (PBMC) from healthy donors and MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Major Multiple Sclerosis (MS) Patients
* RR MS patients without treatment (early stage disease) Or RR MS patients treated with first-line compounds (IFNβ, glatiramer acetate, teriflunomide and dimethyl fumarate, ...).

Or RR MS patients treated with second-line compounds (natalizumab and fingolimod, ...) RR MS patients treated with third-line compounds (alemtuzumab, ...) Or Patients with progressive MS

* Patients who have read and understood the information letter and signed the consent form
* Person affiliated to a social security system

Exclusion Criteria:

* Patients under 18 years of age or over 65 years of age,
* Patients who have benefited from immunosuppressive treatments for other autoimmune or cancerous pathologies,
* Patients receiving treatments for multiple sclerosis and participating in phase 2, 3 or 4 protocols will be excluded.
* Patients who have been treated for less than 1 year with cladribine, daclizumab, ocrelizumab, rituximab will be excluded.
* Patients who have received mitoxantrone or a stem cell transplant,
* Regulatory Criteria :
* Person deprived of liberty by an administrative or judicial decision
* Person placed under legal protection, sub-tutorship or curatorship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-08-13 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Description of cladribine's effects on immune system of multiple sclerosis patients | Through study completion, of 1 year
  Analysis of T cell response by flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France